CLINICAL TRIAL: NCT06647927
Title: Unveiling the Genetic Landscape of Brugada Syndrome: Novel Biomarker Discovery for Precise Diagnosis
Brief Title: GenLab: Unveiling the Genetic Landscape of Brugada Syndrome: Novel Biomarker Discovery for Precise Diagnosis
Acronym: GenLaB
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Azienda Ospedaliero Universitaria di Sassari (Other); The National Research Council, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: PNRR-POC-2023-12378388
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Brugada Syndrome (BrS)
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BrS Affected: The Study population will be composed by patients affected by the Brugada Syndrome, including both the ones already under teatment and subjects with new diagnosis.

SUMMARY:
This research makes several significant contributions to the field of BrS. It employs advanced genetic sequencing techniques to develop a genetic signature to improve the accuracy and efficiency of BrS diagnosis. The identification of specific biomolecular profiles and genetic signatures enhances our understanding of the syndrome's molecular mechanisms, facilitating targeted therapies and refined risk stratification. These advancements optimize patient care by enabling personalized treatment plans and risk assessment. Overall, this research adds value by advancing diagnostic methods, providing molecular insights, optimizing patient care, and positively impacting public health outcomes in BrS.

DETAILED DESCRIPTION:
Our work on BrS is dedicated to decipher the pathogenic mechanism and to ameliorate diagnostic approaches by developing a non-invasive test. Employing a multi-omic strategy, we've identified potential biomarkers across proteins, metabolites, and lipids, leading to a filed patent for a promising biomolecular signature. Additionally, we've discovered associated gene mutations. This grant proposal aims to enhance our preliminary findings by studying a larger BrS cohort, supported by a meticulously curated patient registry. By integrating advanced whole-exome sequencing (WES) and machine learning , we aim to identify a genetic signature for BrS diagnosis and uncover altered pathways integral to BrS etiology. This could refine risk stratification strategies, contributing to improved diagnostic accuracy and deeper understanding BrS molecular mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients affected by Brugada Syndrome
* Patients who signs the Informed Consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 350 patients affected by BrS coming from the same geographical area and age-sex balanced, when it's possible. The total sample includes at least 300 individuals from Sardinia, to whom pre-existing data of 100 patients will be added, already subject to the Whole Exome Sequencing (WES) at Policlinico San Donato.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Multigenic Risk Score (MRS) | from October 2025 to June 2026
  Our objective is to utilize the extensive Whole-Exome Sequencing (WES) data from our cohort to discover shared genetic mechanisms underlying BrS.
  We will conduct rigorous quality control and genome-wide association analyses to identify both common and rare mutations related to BrS. We aim to develop a Multigenic Risk Score (MRS) based on the cumulative findings, considering the effects of associated variants on protein and gene expression levels, and chromatin structure. The MRS seeks to refine the BrS biomarker panel and develop a robust diagnostic tool for BrS by leveraging genetics, machine learning, and translational research.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, Milan, Italy